CLINICAL TRIAL: NCT04682938
Title: The Prevalence and Characteristics of Adrenal Incidentaloma: A Prospective Study
Brief Title: The Prevalence and Characteristics of Adrenal Incidentaloma
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Prof., Chongqing Medical University
Other Study IDs: AI-China2020
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Prevalence; Adrenal Incidentaloma
Keywords: Prevalence; characteristics; adrenal incidentaloma
MeSH Terms: conditions — Adrenal incidentaloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Some subtye of disease should be diagnosed by DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adrenal incidentalomas in Chinese community adults: On weekdays, the first 100 individuals, aged 18 to 78 years, taking health checkup in the Community Health Examination Center were invited to take part in the study.

SUMMARY:
To investige the prevalence, characteristics and prognosis of adrenal incidentalomas in Chinese adults.

DETAILED DESCRIPTION:
With the development of imaging detection technology and its wide application in clinic, the detection rate of adrenal incidentaloma (AI) has been greatly improved. Most AI are benign and do not have the function of autonomic hormone secretion, but about 20% of them have function and can secrete adrenal hormone autonomously. Studies based on biopsy reports show that the prevalence of AI is about 2%, and the prevalence of AI detected by CT scan is 1% - 4.5%. However, most of these studies are retrospective, and there may be selection bias and other confounding factors. There is no large sample prospective study on the prevalence of AI in the general population. The purpose of this study is to prospectively include patients with adrenal incidentaloma in community physical examination population, and evaluate their function and prognosis. The research results will provide new evidence for standardized diagnosis and treatment of adrenal incidentaloma in the future.

ELIGIBILITY:
Inclusion Criteria:

·On weekdays, the first 100 individuals, aged 18 to 78 years, taking health checkup in the Community Health Examination Center were invited to take part in the study.

Exclusion Criteria:

* with known adrenal diseases;
* with continuous steroids or drug treatment that might influence cortisol secretion ordexamethasone metabolism and could not be stopped
* refuse to participate in the study.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese community adults
Sampling Method: Non-Probability Sample
Enrollment: 25356 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence and Characteristics of Adrenal Incidentaloma | 1 years
  To investigate the prevalence and characteristics of Adrenal Incidentaloma in general population in China

SECONDARY OUTCOMES:
Steroid hormones in the function of Adrenal Incidentaloma | 1 years
  prospectively evaluate potential predictive role of combined detection of multiple steroid hormones in the function of Adrenal Incidentaloma

CONTACTS AND LOCATIONS:
Overall Officials: Li Qifu, PhD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, China, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ichijo T, Ueshiba H, Nawata H, Yanase T. A nationwide survey of adrenal incidentalomas in Japan: the first report of clinical and epidemiological features. Endocr J. 2020 Feb 28;67(2):141-152. doi: 10.1507/endocrj.EJ18-0486. Epub 2019 Nov 7. PMID 31694993
- [Result] Lee JM, Kim MK, Ko SH, Koh JM, Kim BY, Kim SW, Kim SK, Kim HJ, Ryu OH, Park J, Lim JS, Kim SY, Shong YK, Yoo SJ; Korean Endocrine Society, Committee for Clinical Practice Guidelines. Clinical Guidelines for the Management of Adrenal Incidentaloma. Endocrinol Metab (Seoul). 2017 Jun;32(2):200-218. doi: 10.3803/EnM.2017.32.2.200. PMID 28685511
- [Result] Fassnacht M, Arlt W, Bancos I, Dralle H, Newell-Price J, Sahdev A, Tabarin A, Terzolo M, Tsagarakis S, Dekkers OM. Management of adrenal incidentalomas: European Society of Endocrinology Clinical Practice Guideline in collaboration with the European Network for the Study of Adrenal Tumors. Eur J Endocrinol. 2016 Aug;175(2):G1-G34. doi: 10.1530/EJE-16-0467. PMID 27390021
- [Derived] Jing Y, Hu J, Luo R, Mao Y, Luo Z, Zhang M, Yang J, Song Y, Feng Z, Wang Z, Cheng Q, Ma L, Yang Y, Zhong L, Du Z, Wang Y, Luo T, He W, Sun Y, Lv F, Li Q, Yang S. Prevalence and Characteristics of Adrenal Tumors in an Unselected Screening Population : A Cross-Sectional Study. Ann Intern Med. 2022 Oct;175(10):1383-1391. doi: 10.7326/M22-1619. Epub 2022 Sep 13. PMID 36095315